CLINICAL TRIAL: NCT06789341
Title: Retrospective Data Collection for a Correlation Study Between Gastric Cancer and Clinical and Laboratory Variables
Acronym: HP-RETROSS
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: HP-RETROSS
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancer Patient
Keywords: gastric cancer, helicobacter pylori
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, retrospective, case-control, single-center, national study that involves the collection of anamnestic, clinical and therapeutic data of patients diagnosed with gastric cancer by histological examination at the Pathological Anatomy Unit (Prof. D'Errico) in the period 2016-2020.

DETAILED DESCRIPTION:
The corresponding medical records will be analyzed to derive information on the socio-demographic characteristics and risk factors of the included subjects. Each case will be paired with two controls chosen from patients who have performed a gastric biopsy with relative histological examination during an endoscopic examination carried out at the IRCCS Azienda Ospedaliero-Universitaria of Bologna.

ELIGIBILITY:
Inclusion Criteria cases:

* Età > 18 anni.
* Diagnosi istologica di carcinoma gastrico
* Ottenimento del consenso informato.

Inclusion criteria controls:

* Età > 18 anni.
* Esecuzione di indagine endoscopica gastrica con relativo esame istologico (mucosa sana, gastrite acuta, gastrite cronica con o senza infezione da Helicobacter pylori, metaplasia intestinale)
* Ottenimento del consenso informato.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Saranno considerati eleggibili ad entrare nella raccolta dati tutti i pazienti con diagnosi di carcinoma gastrico (casi) o che abbiano effettuato un esame istologico gastrico (controlli) rilevati nell'archivio elettronico dell'istituto di anatomia patologica dal 2016 al 2020.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Collection of data | 2016-2020
  The main objective of the study is to create a collection of clinical and laboratory data that will allow us to describe the incidence of gastric cancer in our center and to identify risk factors associated with the disease (H. pylori infection, smoking, alcohol, diet and BMI).

SECONDARY OUTCOMES:
Data interaction in the developement of gastric cancer | 2016-2020
  The secondary objective of the study is to know, analyze and describe the data collected in order to evaluate their possible interaction on the development of gastric neoplastic pathology, and to design a future prospective case-control study.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Fiorini, MD, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No